CLINICAL TRIAL: NCT07085533
Title: Color Vision Loss Progression in IRD Patients: Retinal Structural Changes Correlations, and a Novel Color Discrimination Test for Extreme Low Vision Patients
Brief Title: Natural History Study of Inherited Retinal Diseases
Acronym: MojiLVCDT
Status: Recruiting | Type: Observational
Sponsor: Zhongmou Therapeutics (Industry)
Collaborators: Wuhan University (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: Moji test-01
Record Dates: First submitted 2025-06-03; First posted 2025-07-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-07

CONDITIONS: Retinal Dystrophies; Color Vision Defects; Vision Disorders; Macular Degeneration; Achromatopsia; Optical Coherence Tomography (OCT); Visual Acuity; Genotype; Mutation; Phenotype
Keywords: observational; IRD; ultra low vision; inherited retinal disease; color vision; color test
MeSH Terms: conditions — Retinal Dystrophies; Color Vision Defects; Vision Disorders; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: IRD participants: Individuals in the IRD participants group should have a clinical diagnosis of an inherited retinal dystrophy (such as retinitis pigmentosa, cone or cone-rod dystrophy, rod-cone dystrophy, achromatopsia, etc.). This can be confirmed by genetic testing and comprehensive clinical evaluation ( Best-Corrected Visual Acuity (BCVA), Color Vision Assessment, Visual Field Testing, Full-Field Electroretinography (ffERG), Multifocal ERG (mfERG), Electrooculography (EOG), Optical Coherence Tomography (OCT), Fundus Autofluorescence (FAF), Color Fundus Photography, Dark Adaptometry, Optical Coherence Tomography Angiography (OCTA)).
- Control Group: Non- IRD participants: participants without IRD

SUMMARY:
This prospective, observational investigation seeks to delineate the interplay between chromatic vision deficits and both functional visual outcomes and anatomical retinal biomarkers in individuals affected by Inherited Retinal Dystrophies (IRDs). The study will recruit approximately 200 subjects, encompassing a heterogeneous population of IRD patients-spanning a range of genotypes and clinical severities-as well as control participants devoid of retinal pathology. All enrolled individuals will undergo a standardized battery of evaluations, including quantitative color vision assessment, best-corrected visual acuity (BCVA) determination, and advanced multimodal retinal imaging.

The principal aim is to characterize the relationship between impairments in color discrimination and morphologic disruptions within the outer retinal layers, with particular emphasis on the continuity and reflectivity of the ellipsoid zone (EZ)-historically referred to as the inner segment/outer segment (IS/OS) junction-assessed through spectral-domain optical coherence tomography (SD-OCT). Further, the study will explore associations between chromatic perceptual deficits and underlying genetic mutations, mutation patterns specific to IRD subtypes, and the influence of patient age on the severity and progression of color vision loss.

A key secondary objective is the clinical appraisal and validation of a novel diagnostic modality, the Moji Low-Vision Color Discrimination Test (Moji Test), which is specifically engineered to quantify residual color perception in individuals with advanced central visual impairment. The test's discriminatory capacity will be benchmarked against established color vision testing paradigms to assess its reliability, clinical sensitivity, and suitability for implementation in populations with severe visual acuity reduction.

By incorporating a genetically and phenotypically diverse IRD cohort, the study is designed to enable granular, stratified analyses that will refine the understanding of structural-functional correlations in hereditary retinal disease. The inclusion of a control group with preserved retinal architecture and normal color vision function will provide essential normative baselines for comparative evaluation and statistical inference.

DETAILED DESCRIPTION:
Inherited retinal dystrophies (IRDs) encompass a broad and genetically diverse class of monogenic disorders marked by progressive degeneration of retinal photoreceptors-namely, rods and cones-which ultimately culminates in irreversible visual dysfunction. As the degenerative process advances, patients frequently develop a combination of central and peripheral visual loss alongside progressive impairments in color discrimination. Among retinal structural biomarkers, the ellipsoid zone (EZ)-a hyperreflective band corresponding to the mitochondria-dense segment of the photoreceptor inner segments, historically denoted as the IS/OS junction in spectral-domain optical coherence tomography (SD-OCT)-has emerged as a key indicator of residual photoreceptor viability and visual function. Prior studies, particularly those focusing on retinitis pigmentosa (RP), have demonstrated a compelling association between EZ integrity and chromatic discrimination ability, reinforcing the critical relationship between anatomical preservation and functional outcomes in retinal dystrophies.

This prospective investigation is designed to quantitatively characterize color vision performance in individuals with IRDs and to evaluate its association with retinal microstructural features as revealed by multimodal imaging modalities, including SD-OCT-derived EZ measurements, total retinal thickness, and best-corrected visual acuity (BCVA). By integrating these anatomical measures with genotypic data, the study will further examine the influence of specific mutation types, allelic patterns, and patient age on chromatic function, thereby offering a comprehensive analysis of genotype-phenotype relationships in IRD-associated dyschromatopsia.

A persistent challenge in the evaluation of color vision among IRD patients-particularly those with advanced vision loss-is the limited applicability of conventional color vision assessments. Standard psychophysical tests, such as the Ishihara pseudoisochromatic plates and the Farnsworth-Munsell 100 Hue Test, are fundamentally dependent on preserved spatial resolution and pattern recognition, thereby rendering them ineffective in individuals with substantial visual acuity deficits. Although the Low Vision Cambridge Color Test (lvCCT) offers a more accessible alternative for patients with moderate acuity impairment, those with BCVA at or below the level of Counting Fingers (logMAR ≥ 1.6) are frequently unable to complete the test, resulting in inconclusive or misleading data regarding true chromatic capability. In such cases, performance failure often reflects the constraints of visual resolution rather than an authentic deficit in color discrimination, complicating both diagnosis and longitudinal monitoring.

To address these limitations, the present study incorporates the Moji Low-Vision Color Discrimination Test (Moji LVCDT)-a novel chromatic assessment tool specifically developed for individuals with profound visual impairment. This test employs high-contrast, large-format color stimuli, enabling the assessment of chromatic discrimination thresholds independent of fine spatial vision. Preliminary validation data indicate that the Moji LVCDT can successfully detect residual color perception in patients who are unable to engage with standard color vision testing paradigms, thereby providing clinically meaningful results even in the most advanced stages of IRD.

As part of the study protocol, the Moji LVCDT will be administered in parallel with established color vision tests, including the Ishihara plates and the low-vision-adapted Cambridge Color Test, to evaluate its diagnostic sensitivity, specificity, and correlation with both functional vision and structural retinal metrics. Through comparative analysis, the study aims to validate the Moji LVCDT as a reliable and scalable tool for quantifying color vision in populations historically excluded from color function assessments due to visual acuity constraints.

By integrating structural, functional, and genetic data, this investigation seeks to advance current understanding of the pathophysiological basis of color vision loss in inherited retinal diseases. Moreover, the validation of the Moji LVCDT may lay the foundation for the establishment of a standardized, clinically applicable method for tracking chromatic function in low-vision populations. The outcomes of this study have the potential to enhance diagnostic precision, inform clinical management strategies, and provide a sensitive outcome measure for use in future interventional trials targeting retinal preservation and visual function restoration in IRD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Color Perception and Communication Ability Participants must have the ability to verbally identify or describe colors and test stimuli. This requires adequate cognitive and communicative capacity to understand instructions and respond appropriately during color vision testing.
2. Diagnosis of Inherited Retinal Dystrophy (IRD Group Only) Participants assigned to the IRD group must have a confirmed clinical diagnosis of an inherited retinal dystrophy
3. No Evidence of Inherited Retinal Disease (Control Group Only)

Participants in the control group must have:

* No known history or clinical evidence of inherited retinal degeneration
* Normal retinal health or only non-retinal ocular conditions not affecting retinal function (e.g., mild cataract, corrected refractive error)
* Normal or expected-normal color vision

Exclusion Criteria:

1. Non retinal causes of color vision loss

   * Optic neuropathies (e.g., optic neuritis, glaucoma related optic nerve damage)
   * Cortical vision impairments affecting color perception
   * Any other neurological or optic nerve pathology causing color vision deficiency
2. Psychological or cognitive conditions affecting color perception or communication

   * Severe developmental delays
   * Cognitive impairments interfering with ability to comprehend or reliably perform color vision tests
   * Psychiatric conditions that impair visual interpretation or reliable testing
3. Prior treatment with potential transient effects on the retina

   * Recent retinal surgery
   * Recent drug therapy affecting retinal structure or function
   * Any acute intervention that might confound the correlation analyses due to lack of a stable baseline

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with inherited retinal diseases (IRD) and non-IRD individuals
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2027-06-04 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Moji Low Vision Color Discrimination Test with other color discrimination tests in detecting participants' color vision ability. | Baseline (single visit)
  Color vision ability will be measured by three different color discrimination tests including Ishihara color test, Low Vision Cambridge Color test (LVCCT), and Moji Low vision Color Discrimination Test (Moji LVCDT). The result will be presented as the score/full score (unit: %) for each test. And the respond percentage of the participants for each test will be compared.
Evaluating the efficiency of Moji LVCDT in participants with extreme Low BCVA | Baseline (single visit)
  Moji LVCDT is conducted using novel Moji test device and protocol to detect the color vision ability of participants. This test can be performed for participants with best corrected visual acuity (BCVA) from normal vision to participants with light perception BCVA, focusing whether having the best efficiency for the participants with extreme low vision (LogMAR 1.6 and above).

SECONDARY OUTCOMES:
Evaluating the correlation Between Color Vision Loss (unit: Ishihara color test result score percentage) and IS/OS junction length (unit: μm). | Baseline (single visit)
  Retinal structural changes assessed by measuring the structural changes in optic coherence tomography (OCT) (IS/OS junction length, unit: μm) and obtained score in Ishihara color test (unit: Ishihara color test result score percentage).
Evaluating the correlation Between Color Vision Loss (unit: Low Vision Cambridge Color Vision Test result score percentage) and IS/OS junction length (unit: μm). | Baseline (single visit)
  Retinal structural changes assessed by measuring the structural changes in optic coherence tomography (OCT) (IS/OS junction length, unit: μm) and obtained score in Low Vision Cambridge Color Test (unit: Ishihara color test result score percentage).
Evaluating the correlation Between Color Vision Loss (unit: Moji Low Vision Color Discrimination Test result score percentage) and IS/OS junction length (unit: μm). | Baseline (single visit)
  Retinal structural changes assessed by measuring the structural changes in optic coherence tomography (OCT) (IS/OS junction length, unit: μm) and obtained score in Moji Low Vision Color Discrimination Test (unit: Ishihara color test result score percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Yin Shen, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, China

IPD SHARING:
Plan to Share IPD: Undecided